CLINICAL TRIAL: NCT06861465
Title: EMPower Mechanisms: an Evidence-based Mental Wellness Programming Online for People with Primary Biliary Cholangitis - a Feasibility Randomized Controlled Trial
Brief Title: EMPower Mechanisms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Puneeta Tandon, Associate Professor, Principal Investigator, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00144631
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Primary Biliary Cholangitis (PBC)
Keywords: Mind Body Wellness; Quality of Life; Fatigue; Cognitive Function; Physical Function; Mental Health
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Fatigue; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Online Mind-Body Program (Active Comparator): Online program (mindful movement, meditation, breathwork)
  Interventions: Behavioral: Online Mind-Body Wellness Program
- Experimental: Online Mind-Body Program + Nutritional Counselling (Experimental): Online program (mindful movement, meditation, breathwork) + nutritional counselling
  Interventions: Behavioral: Online Mind-Body Wellness Program + Nutritional Counselling

INTERVENTIONS:
Behavioral: Online Mind-Body Wellness Program — Online program (mindful movement, meditation, breathwork)
  Arms: Experimental: Online Mind-Body Program
Behavioral: Online Mind-Body Wellness Program + Nutritional Counselling — Online program (mindful movement, meditation, breathwork) + nutrition counselling
  Arms: Experimental: Online Mind-Body Program + Nutritional Counselling

SUMMARY:
Primary Biliary Cholangitis (PBC) is a chronic liver disease that can cause fatigue, itching, brain fog, and emotional distress, all of which can lower quality of life. While the standard treatment, ursodeoxycholic acid (UDCA), helps slow the disease, it does not relieve these symptoms. Research shows that mind-body practices-such as breathing exercises, meditation, and gentle movement-can help improve mental and physical well-being in people with chronic conditions, but their benefits for PBC are not yet well understood.

This study will test a 10-week online wellness program designed for women with PBC. The program will include guided breathing, meditation, and movement exercises, plus optional weekly group sessions and educational videos. Some participants will also receive nutrition guidance on the Mediterranean diet to see if it adds extra benefits.

The study will evaluate feasibility via recruitment, adherence, and retention. To assess acceptability, participants will provide feedback through surveys and interviews. The study will also explore early signs of effectiveness by measuring changes in symptoms like anxiety, depression, fatigue, and stress, as well as biological markers, brain activity, physical function, and data from wearable devices.

The results will help determine whether an online mind-body program, with or without nutrition support, could be a simple and effective way to help people with PBC manage their symptoms and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Primary Biliary Cholangitis (PBC) as confirmed by a study Hepatologist using accepted clinical criteria
* Have been on stable medical therapy for PBC for ≥3 months
* Score ≥3 on a 1-10 numeric rating scale for two of: depression, anxiety, fatigue, sleep disturbance, cognitive impairment
* Are able to communicate in English
* Have access to an Internet-connected device in their home
* Can commit to up to 60 minutes of study activities 5 days per week

Exclusion Criteria:

* Unable to provide informed consent
* Have decompensated cirrhosis including hepatic encephalopathy
* Are post-liver transplant
* Current severe substance use or psychiatric disorder judged to interfere with study testing or program participation
* Are receiving compassionate care
* Have a clinical condition that makes the intervention unsafe or infeasible (e.g. unable to follow instruction) or unsafe environment for virtual participation
* Practices mind-body practices more than the study dose
* Have contraindications for MRI
* Have colour blindness
* Are unable to attend baseline testing

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Intervention | Baseline and Week 10
  Feasibility will be assessed by (i) adherence rate (percentage completing ≥70% of intervention, target ≥70%), and (ii) retention rate (percentage completing baseline and follow-up assessments, target ≥70%).
Acceptability of the Intervention | Baseline and Week 10
  Acceptability will be assessed via participant-reported satisfaction with the intervention using numerical surveys and perceived burden of study measures.

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Baseline and Week 10
  Description: Depression and anxiety will be measured on the Hospital Anxiety and Depression Scale. The minimum value is 0, the maximum is 21, and higher scores mean a worse outcome.
Modified Fatigue Impact Scale (MFIS) | Baseline and Week 10
  The Modified Fatigue Impact Scale (MFIS) assesses the effect of fatigue on cognitive functioning, physical functioning, and psychosocial functioning. The minimum value is 0, the maximum value is 84, and higher scores mean a worse outcome.
Primary Biliary Cholangitis-40 (PBC-40) | Baseline and Week 10
  The PBC-40 assesses quality of life (HRQoL) in individuals with PBC. It consists of 40 items across six domains, assessing symptoms, fatigue, emotional well-being, cognitive function, social impact, and itch.
Perceived Stress Scale (PSS) | Baseline and Week 10
  The Perceived Stress Scale (PSS) assesses how unpredictable, uncontrollable, and overwhelming individuals find their lives. The scale is scored from 0 to 40. Higher scores indicate greater perceived stress.
Sleep Disturbance | Baseline and Week 10
  Sleep disturbance will be measured using the PROMIS Sleep Disturbance 6a. The scale ranges from 8 to 40. Higher scores indicate greater sleep disturbance.
Cognitive Function | Baseline and Week 10
  The PROMIS Short Form - Cognitive Function 6a will be used to assess cognitive function. The scale measures self-reported cognitive function on a scale from 6 to 30. Higher scores indicate better cognitive function.
Pain Interference | Baseline and Week 10
  Pain interference will be measured using the PROMIS Short Form - Pain Interference 4a. The measure assesses the impact of pain on daily activities on a scale from 4 to 20. Higher scores indicate greater pain interference.
Itch Interference | Baseline and Week 10
  Itch interference will be measured using the The PROMIS Short Form - Itch Interference 4a. The measure assesses the impact of itching on daily activities on a scale from 4 to 20. Higher scores indicate greater itch interference.
Changes in Biological Markers | Baseline and Week 10
  Blood sample analysis for biomarkers related to stress and inflammation
  Measure: Levels of stress, inflammation, and fatigue biomarkers (e.g., cortisol, cytokines)
Neurophysiological Changes | Baseline and Week 10
  Pre-post intervention changes in brain activity patterns
  Measure: fMRI and fNIRS measures of brain function
Sit-to-stand | Baseline and Week 10
  The Sit-to-Stand Test measures lower body strength and functional mobility by assessing the number of times an individual can rise from a seated position to a standing position within a set time or the time taken to complete a set number of repetitions. Higher repetitions in a given time or a shorter completion time indicate better functional performance.
The 2-Minute Step Test (2MST) | Baseline and Week 10
  The 2-Minute Step Test (2MST) measures aerobic endurance by counting the number of steps a person takes in place within 2 minutes, lifting the knees to a standardized height. Higher step counts indicate better endurance and functional fitness.
Changes in Exercise Tolerance Mechanisms | Baseline and Week 10
  Assessed using physiological testing for exercise tolerance.
  Measures: Non-invasive estimates of pulmonary oxygen uptake, skeletal muscle oxygenation
Changes in Wearable-Based Measures | Baseline and Week 10
  Collected via wearable devices to assess cardiovascular function.
  Measure: Heart rate variability
Change in Mediterranean diet score | Baseline and Week 10
  Assessed using dietary recall and adherence questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada